CLINICAL TRIAL: NCT01697943
Title: A Pilot Randomized Controlled Trial Examining the Differences of Quality of Life of Roux-En-Y Pouch Reconstruction and Conventional Roux-En-Y Reconstruction in Patients Undergoing Total Gastrectomy.
Brief Title: Impact of Roux-En-Y Pouch Reconstruction Compared With Conventional Roux-En-Y Reconstruction on Quality of Life in Patients Undergoing Total Gastrectomy
Acronym: GCQOL02
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yanong Wang, Director of Department of Abdominal Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-44-563
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Gastric Tumor
Keywords: Gastric Malignant Tumor; Total Gastrectomy; Reconstruction
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Roux-En-Y Pouch Reconstruction or Roux-En-Y Reconstruction (Experimental)
  Interventions: Procedure: Roux-En-Y Pouch Reconstruction or Conventional Roux-En-Y Reconstruction

INTERVENTIONS:
Procedure: Roux-En-Y Pouch Reconstruction or Conventional Roux-En-Y Reconstruction

SUMMARY:
The purpose of this study is to find out more about differences of the quality of life in patients undergoing Roux-En-Y pouch reconstruction and conventional Roux-En-Y reconstruction. To find a better reconstruction for patients who received total gastrectomy.

DETAILED DESCRIPTION:
Total gastrectomy has been indicated mainly for advanced gastric cancer located from the upper to middle third of the stomach or multiple gastric cancers.The most common method of creating a way for food is called a "Roux-en-Y", in which one part of the intestines is connected with the end of the esophagus (the swallowing tube) in the abdomen, and another connection is made between the intestines ' lower down.

Patients with total gastrectomy suffer from poor food intake, anemia, and poor digestion because of loss of gastric reservoir or a lack of normal hormonal secretion for digestion. It often is associated with a limitation of postoperative quality of life (QOL). To improve postoperative nutritional status and QOL, surgeons have tried to establish ideal reconstruction after total gastrectomy and the optimum procedure for reconstruction has been discussed.

This study will compare the postoperative quality of life (QOL) of gastric pouch reconstruction with the usual reconstruction to see if the pouch makes patients feel better.

ELIGIBILITY:
Inclusion Criteria:

* • Pathologically confirmed gastric malignant tumor at fUSCC (biopsy may be performed at other institutions but slides must be confirmed at SHCA, as is routine care at our institution) , and the patients be assessed must be carried out total gastrectomy by three specialists.

  * Patients 20-75 years old
  * Normal organ function, able to tolerate surgery, no clear contraindication for surgery
  * No evidence of metastases of adjacent organs
  * be able to provide follow-up over 2 years
  * No specific treatment for gastric cancer before surgery
  * In line with the Declaration of Helsinki and the requirements of the hospital ethics committee.
  * The subjects were able to understand and comply with the trial protocol, and signed informed consent.

Exclusion Criteria:

* • Synchronous or metachronous (less than five years) and with other malignancies.

  * Cirrhosis and portal hypertension
  * Associated with blood diseases
  * Serious heart/ lung and kidney dysfunction or with metabolic diseases such as diabetes, hyperthyroidism.
  * Suffering from a serious neurological diseases or psychological diseases affecting the life

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in QOL (Quality of Life) | 5years
  From preoperative following total gastrectomy, as measured with the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 and QLQ-STO22 questionnaires

SECONDARY OUTCOMES:
Nutritional status of patients | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China